CLINICAL TRIAL: NCT00000634
Title: A Pilot Pharmacokinetic Phase I Evaluation of BI-RG-587 in HIV-Infected Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Boehringer Ingelheim (Industry)
Purpose: Treatment
Other Study IDs: ACTG 165; 00853
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2011-03-01 (Estimated); Status verified 2011-02

CONDITIONS: HIV Infections
Keywords: Benzodiazepines; Drug Evaluation; Drugs, Investigational; Acquired Immunodeficiency Syndrome; Antiviral Agents
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Nevirapine

INTERVENTIONS:
Drug: Nevirapine

SUMMARY:
To generate initial information on the pharmacokinetics (blood levels) and dose proportionality of nevirapine (BI-RG-587) plasma levels in HIV-infected children; to assess the safety and tolerance of single rising oral doses of nevirapine in HIV-infected children; and to confirm that the single doses that achieve certain plasma levels in adults achieve similar levels in HIV-infected children.

Test tube studies have shown that nevirapine (BI-RG-587) inhibits replication (reproduction) of HIV. Nevirapine works with zidovudine (AZT) and is active against strains of the virus that are resistant to AZT. Studies of the drug in HIV-infected adults showed no serious adverse effects.

DETAILED DESCRIPTION:
Test tube studies have shown that nevirapine (BI-RG-587) inhibits replication (reproduction) of HIV. Nevirapine works with zidovudine (AZT) and is active against strains of the virus that are resistant to AZT. Studies of the drug in HIV-infected adults showed no serious adverse effects.

Two doses, given by mouth, are evaluated: Three patients receive the lower dose, and 7 days after the third patient receives the lower dose, three additional patients receive the higher dose. After dosing, blood is drawn at 1, 2, 4, 8, 24, 48, 96, 168 hours to measure blood levels of the drug.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Intravenous gammaglobulin. Pneumocystis prophylaxis according to published guidelines.

Patients must have the following:

* HIV infection.
* Parent or guardian must be available to give written informed consent.

Exclusion Criteria

Concurrent Medication:

Excluded:

* Zidovudine (AZT).
* Steroid dependency.

Excluded within 1 hour before and 4 hours after study drug administration:

* Drugs that might interfere with the absorption of study drug (H2 blockers, antacids, carafate, cholestyramine).
* Benzodiazepines.
* Alcohol-containing substances.

Concurrent Treatment:

Excluded:

* Requiring supplemental oxygen.

Patients with the following are excluded:

* Active opportunistic or serious bacterial infection.
* Lymphoid interstitial pneumonitis (LIP) and steroid dependent or requiring supplemental oxygen or have a pretreatment pa02 < 70 mm Hg.
* Pre-existing malignancies.

Prior Medication:

Excluded:

* Zidovudine (AZT) within 7 days prior to administration of study drug.

Excluded for at least 4 weeks prior to drug administration:

* Other approved or investigational antiretroviral agents. All other investigational agents. Biologic response modifiers (e.g., interferon) or immunomodulators. Immunosuppressive agents (including glucocorticoids). Coumadin and other anticoagulant medications.

Prior Treatment:

Excluded:

* Red blood cell transfusion within 4 weeks of study entry.

Patients may not have the following:

* Opportunistic or serious bacterial infection.

Zidovudine (AZT) > 7 days prior to administration of study drug.

Active alcohol or drug abuse.

Ages: 2 Months to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6
Dates: Primary Completion 1995-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Univ of Massachusetts Med Ctr / Biotech II, Worcester, Massachusetts, United States

REFERENCES:
- [Background] Luzuriaga K, Bryson Y, McSherry G, Robinson J, Stechenberg B, Scott G, Lamson M, Cort S, Sullivan JL. Pharmacokinetics, safety, and activity of nevirapine in human immunodeficiency virus type 1-infected children. J Infect Dis. 1996 Oct;174(4):713-21. doi: 10.1093/infdis/174.4.713. PMID 8843207